CLINICAL TRIAL: NCT07321782
Title: Mayer Rokitansky Kuster Hauser (MRKH) Syndrome: A Monocentric Ambispective Study on Clinical and Ultrasound Findings and Novel Imaging-Based Classification
Brief Title: Clinical and Imaging Features in MRKH Syndrome
Acronym: ROK-US
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 8153
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Mayer Rokitansky Kuster Hauser Syndrome; Müllerian Agenesis
MeSH Terms: conditions — Mullerian aplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mayer-Rokitansky-Küster-Hauser (MRKH) syndrome is a congenital condition characterized by uterovaginal agenesis in phenotypically normal women with a 46,XX karyotype. Despite increasing knowledge of its clinical and genetic features, MRKH syndrome shows marked phenotypic heterogeneity, and current classification systems do not fully reflect the wide spectrum of anatomical presentations encountered in clinical practice.

This ambispective, observational, monocenter study aims to describe the clinical, sonographic, radiological, and genetic characteristics of patients with suspected or confirmed MRKH syndrome referred to a tertiary referral center. All enrolled patients will undergo standardized pelvic ultrasound evaluation, including transabdominal and transrectal approaches, with optional MRI according to clinical indications. Sonovaginography will be performed to objectively assess vaginal length. Genetic investigations, including array CGH and next-generation sequencing, will be conducted as part of routine clinical care.

The primary objective is to characterize the clinical and ultrasound features of MRKH syndrome. Secondary objectives include the development of a novel image-based classification system to better describe disease severity and morphological patterns, validation of sonovaginography for vaginal length measurement, and correlation of genetic alterations with ultrasound-based staging. The study aims to improve diagnostic standardization and contribute to a better understanding of the genotype-phenotype relationship in MRKH syndrome.

ELIGIBILITY:
Inclusion Criteria

* Female patients with suspected or previously diagnosed MRKH syndrome
* 46,XX karyotype
* Age 10-60 years
* For prospective patients: signed Informed Consent and Consent to Data Processing (by patient or parent/guardian if minor)
* For retrospective patients: availability of data collected in compliance with Data Protection regulations (DPIA conducted)

Exclusion Criteria

* Patients with other causes of primary amenorrhea (e.g., Androgen Insensitivity Syndrome / Morris syndrome)
* Karyotype different from 46,XX
* For prospective patients: inability to provide informed consent or parental/guardian consent if minor

Ages: 10 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: The study will include female patients aged 10 to 60 years with suspected or previously diagnosed Mayer-Rokitansky-Küster-Hauser (MRKH) syndrome, confirmed by a 46,XX karyotype. Both retrospective and prospective patients referred to the 'Female Genital Tract Anomalies' outpatient clinic at the Department of Obstetrics and Gynecology, IRCCS Fondazione Policlinico Universitario Agostino Gemelli, Rome, Italy, will be included. Prospective participants will provide informed consent (or parental/guardian consent for minors). Retrospective participants will be included based on previously collected data in compliance with data protection regulations. Patients with other causes of primary amenorrhea or non-46,XX karyotype will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Clinical and ultrasonographic characterization of MRKH syndrome | Baseline (at enrollment)
  Description of clinical features and standardized ultrasound findings in patients with Mayer-Rokitansky-Küster-Hauser syndrome, including presence and morphology of uterine remnants, vaginal length, ovarian position and morphology, and associated pelvic or renal anomalies, assessed by transabdominal and transrectal ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Carla Testa, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy